CLINICAL TRIAL: NCT00049179
Title: A Phase II Study of Gemtuzumab Ozogamicin (Mylotarg) and Standard Dose ARA-C for Patients With Relapsed Acute Myeloid Leukemia (AML)
Brief Title: S0117 Gemtuzumab Ozogamicin Plus Cytarabine in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0117; S0117 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Cytarabine; Gemtuzumab

INTERVENTIONS:
Drug: cytarabine — ind and consol: 200 mg/m2/d continuous IV days 1-7
Drug: gemtuzumab ozogamicin — ind and consol: 6 mg/m2 IV over 2 hrs day 1, 4mg/m2 IV over 2 hrs day 8

SUMMARY:
RATIONALE: Monoclonal antibodies such as gemtuzumab ozogamicin can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy such as cytarabine use different ways to stop cancer cells from dividing so they stop growing or die. Combining gemtuzumab ozogamicin with cytarabine may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemtuzumab ozogamicin with cytarabine in treating patients who have relapsed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of gemtuzumab ozogamicin and cytarabine in patients with relapsed acute myeloid leukemia.
* Determine the frequency and severity of toxic effects of this regimen in CD33-positive patients.
* Determine, preliminarily, the prognostic significance of drug resistance phenotype, cytogenetics, and molecular genetic characteristics of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction: Patients receive gemtuzumab ozogamicin IV over at least 2 hours on days 1 and 8 and cytarabine IV continuously over days 1-7.
* Consolidation: Beginning between days 28 and 75, patients who achieve A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status receive one course of gemtuzumab ozogamicin and cisplatin as in induction chemotherapy.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 30-55 patients will be accrued for this study within 10-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia (AML)

  * FAB M1-2 or M4-7
  * No blastic transformation of chronic myelogenous leukemia
* In first relapse after prior complete response

  * Patients who relapsed after autologous or allogeneic bone marrow or peripheral blood stem cell transplantation are not eligible
* CD33 positive
* Prior myelodysplastic syndromes or secondary AML allowed
* Concurrent enrollment on SWOG-9007 (cytogenetics protocol)
* No clinical or documented CNS involvement with AML

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC no greater than 30,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 1.5 times ULN

Renal

* Not specified

Cardiovascular

* No unstable cardiac arrhythmias
* No unstable angina

Other

* HIV negative
* No other malignancy within the past 5 years except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Adequately treated stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior gemtuzumab ozogamicin for AML

Chemotherapy

* Prior hydroxyurea to control high cell counts allowed

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 4 weeks since prior investigational agents and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-04; Primary Completion 2005-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
CR | After induction therapy is completed

CONTACTS AND LOCATIONS:
Overall Officials: John E. Godwin, MD, MS, Study Chair — Loyola University
Locations (151):
- United States (151):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Mills-Peninsula Health Services, Burlingame, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center at Stormont-Vail Regional Health Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Cancer Center at Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Orange Regional Medical Center - Horton Campus, Middletown, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Cancer Care Center at Skagit Valley Hospital, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Center at Southwest Washington Medical Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Welch Cancer Center, Sheridan, Wyoming